CLINICAL TRIAL: NCT05994092
Title: Influence of Voluntary Isocapnic Hyperpnea on Blood Lactate Level and Rate of Perceived Exertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Sport - National Research Institute, Poland (Other)
Responsible Party: Principal Investigator, Tomasz Kowalski, Principal Investigator, Institute of Sport - National Research Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TK03/2023
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Blood Lactate Decrease
Keywords: Voluntary Isocapnic Hyperpnea; Lactate Clearance

STUDY DESIGN:
Intervention Model Description: Parallel Group Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: Voluntary Isocapnic Hyperpnea
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Voluntary Isocapnic Hyperpnea — The protocol of 3' of breathing with 20 breaths·min-1 frequency. The Isocapnic BreathWayBetter devices (Isocapnic Technologies Inc, Kelowna, Canada) with 6-liter bags were used. The protocol was performed in a seating position.
  Arms: Experimental

SUMMARY:
All the study participants performed the Wingate Anaerobic Test (WAnT) with maximal effort. The experimental group (E) performed a 3-minute recovery protocol based on low-intensity breathing Voluntary Isocapnic Hyperpnea exercises 20 minuter after cessation of the exercise, whereas the control group (C) used passive recovery only. All study participants were advised to sit during the 30-minute period, with minimal walking in order to meet the physiological needs allowed. The blood samples were taken 3 minutes and 30 minutes after cessation of the exercise to measure the bLa. The Borg CR-10 Scale was presented to the participants 3 minutes and 30 minutes after cessation of the exercise to measure the rate of perceived exertion (RPE) (Borg, 1998).

DETAILED DESCRIPTION:
All the study participants performed the Wingate Anaerobic Test (WAnT) with maximal effort. The experimental group (E) performed a 3-minute recovery protocol based on low-intensity breathing VIH exercises 20 minuter after cessation of the exercise, whereas the control group (C) used passive recovery only. All study participants were advised to sit during the 30-minute period, with minimal walking in order to meet the physiological needs allowed. The blood samples were taken 3 minutes and 30 minutes after cessation of the exercise to measure the bLa. The Borg CR-10 Scale was presented to the participants 3 minutes and 30 minutes after cessation of the exercise to measure the rate of perceived exertion (RPE).

WAnT was conducted using a Monark 874E Cycle Ergometer (Monark Exercise AB, Sweden). Prior to the test, a standard warm-up of 5 minutes was performed with a load of 0.8-1.2 W/kg. Then, athletes performed a maximal 6-second sprint with a load adjusted to 7.5% of the individual body weight. Following a 2-minute rest period, the athletes underwent a 30-second WAnT with the load adjusted to 7.5% of the individual body weight. The objective for the subjects was to achieve the highest possible peak power as fast as possible and maintain the highest power output throughout the whole test duration. Loud and dynamic verbal encouragement was provided. The testing took place between 9:00 and 10:30 AM. The basic mechanical parameters of the exercise, including performed work and maximum power, were computed with dedicated software (MCE 6.0 - JBA Z. Staniak, Poland) linked to the cycle ergometer.

The recovery protocol consisted of 3' of breathing with 20 breaths·min-1 frequency. The Isocapnic BreathWayBetter devices (Isocapnic Technologies Inc, Kelowna, Canada) with 6-liter bags were used. The protocol was performed in a seating position.

Blood samples were taken from fingertips by skilled technicians to 20 uL capillary tubes. bLa was measured with Super GL2 analyzer (Dr. Müller Gerätebau GmbH, Freital, Germany).

Whereas participants and data collectors were aware of the allocated training method, the laboratory technicians performing biochemistry assays were kept blinded to the allocation. The participants were assigned at random to either E or C group to perform VIH protocol under a supervision of qualified physiotherapist.

Stratified randomization to assign the participants was used. First, the participants were assigned to subgroups based on the membership in National Development or National Elite Team. Then, the participants were assigned to subgroups based on the gender. Then, the participants were assigned to E or C group based on the coin toss.

ELIGIBILITY:
The inclusion criteria:

* valid medical certificate to compete in speedskating,
* lack of previous experience with RMT,
* at least 6 years of athletic training.

The exclusion criteria:

* any chronic medical condition,
* any acute medical condition within last 3 months,
* any ongoing medication intake.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in blood lactate (bLa) | 30 minutes
  The blood samples were taken 3 minutes and 30 minutes after cessation of the exercise to measure the bLa.
  Blood samples were taken from fingertips by skilled technicians to 20 uL capillary tubes. bLa was measured with Super GL2 analyzer (Dr. Müller Gerätebau GmbH, Freital, Germany).
Changes in rate of perceived exertion (RPE) | 30 minutes
  The Borg CR-10 Scale was presented to the participants 3 minutes and 30 minutes after cessation of the exercise to measure the rate of perceived exertion (RPE) (Borg, 1998).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sport - National Research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request.

REFERENCES:
- [Derived] Kowalski T, Wilk A, Rebis K, Lohse KM, Sadowska D, Klusiewicz A. Influence of voluntary isocapnic hyperpnoea on recovery after high-intensity exercise in elite short-track speedskaters - randomized controlled trial. BMC Sports Sci Med Rehabil. 2024 Jun 20;16(1):137. doi: 10.1186/s13102-024-00927-0. PMID 38902811